CLINICAL TRIAL: NCT01133210
Title: Effect of Maraviroc on Metabolic Function in Obese Subjects (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0533
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; triglyceride; cholesterol; Maraviroc
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Experimental): Subjects will receive 12 weeks of treatment with maraviroc (300 mg po bid).
  Interventions: Drug: Maraviroc
- Placebo (Placebo Comparator): Subjects will receive 12 weeks of treatment with placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Maraviroc — dosage will be a 300mg Maraviroc pill twice a day for 12 weeks
  Other Names: Selzentry; Celsentri
  Arms: Maraviroc
Other: placebo — subjects will be given placebo pills with instructions to take one pill twice a day for 12 weeks.
  Other Names: control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of maraviroc therapy in obese insulin resistant subjects on:

1. Plasma triglyceride concentration
2. Plasma HDL-cholesterol and LDL-cholesterol concentrations
3. Plasma markers of cardiometabolic risk and inflammation

DETAILED DESCRIPTION:
The purpose of this study is to determine, in obese insulin resistant subjects, the effect of maraviroc therapy, a selective antagonist of the human chemokine receptor CCR5, on:

1. Plasma triglyceride concentration
2. Plasma HDL-cholesterol and LDL-cholesterol concentrations
3. Plasma markers of cardiometabolic risk and inflammation

ELIGIBILITY:
Inclusion Criteria:

* obese (body mass index (BMI) between 30 and 45.9)
* increased plasma triglyceride concentrations (150-400 mg/dL)

Exclusion Criteria:

* active or previous infection with hepatitis B or C
* history of alcohol abuse
* current alcohol consumption (>20g/day)
* severe hypertriglyceridemia (>400 mg/dL)
* active peptic ulcer disease
* diabetes
* pregnant or lactating
* take statins, fibrates, niacin, moderate to strong Cyp3A4 inhibitors or inducers, or any other medication that might confound interpretation of the study results will be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
effect of Maraviroc on plasma triglyceride concentration | 12 weeks
  We will compare pre and post-treatment serum triglyceride concentrations in subjects receiving a 12 week course of either Maraviroc or placebo.

SECONDARY OUTCOMES:
Effect of Maraviroc on serum HDL concentration | 12 weeks
  We will compare pre and post-treatment serum HDL concentrations in subjects receiving a 12 week course of either Maraviroc or placebo.
effect of Maraviroc on serum LDL-cholesterol concentration | 12 weeks
  We will compare pre and post-treatment serum LDL-cholesterol concentrations in subjects receiving a 12 week course of either Maraviroc or placebo.
Effect of Maraviroc on plasma markers of cardiometabolic risk and inflammation | 12 weeks
  We will compare pre and post-treatment plasma concentrations of C-reactive protein and InterLeukin-6 in subjects receiving a 12 week course of either Maraviroc or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States